CLINICAL TRIAL: NCT06598267
Title: A Prospective,Single-center,Randomized,Controlled Study to Evaluate the Efficacy and Safety of SASI Compared with RYGB in the Treatment of Obesity and Related Metabolic Diseases
Brief Title: Evaluate the Efficacy and Safety of SASI Compared with RYGB in the Treatment of Obesity and Related Metabolic Diseases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Xuehui Chu, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-557
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Bariatric Surgery
Keywords: Obesity and Related Metabolic Disease
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SASI group (Experimental): single anastomosis sleeve ileal bypass
  Interventions: Procedure: SASI
- RYGB group (Experimental): Roux-en-Y gastric bypass
  Interventions: Procedure: RYGB

INTERVENTIONS:
Procedure: SASI — single anastomosis sleeve ileal bypass
  Arms: SASI group
Procedure: RYGB — Roux-en-Y gastric bypass
  Arms: RYGB group

SUMMARY:
Single anastomosis sleeve ileal bypass (SASI) is an improved surgical technique for sleeve gastrectomy (SG), which combines the advantages of SG and Roux-en-Y gastric bypass (RYGB) while avoiding their disadvantages,in order to achieve better treatment outcomes.On the one hand,SASI surgery improves the effectiveness of weight loss surgery by adding gastrointestinal anastomosis on the basis of SG,while reducing gastric pressure and improving postoperative gastroesophageal reflux symptoms.On the other hand,it also avoids the regret of RYGB surgery leaving the stomach open for gastroscopy examination and reduces the risk of postoperative nutrition related complications.Therefore,SASI surgery has demonstrated good application prospects and is expected to be promoted in clinical practice.So far,there has been no comparative study of RCTs between RYGB and SASI internationally.In order to compare the weight loss effects of SASI and RYGB surgery,this study intends to conduct a randomized controlled trial on patients who meet the criteria and require weight loss surgery,providing high-level evidence-based medicine for the further clinical development of SASI surgery in the future.

DETAILED DESCRIPTION:
Routine preoperative examinations should be conducted on patients planning to undergo weight loss surgery,and inclusion screening should be conducted according to the inclusion and exclusion criteria.Patients who meet the inclusion criteria will receive informed consent before enrollment and be randomly assigned to either the experimental group (SASI group) or the control group (RYGB group) for weight loss surgery based on computer randomization results.

Monitor the patient's surgical condition and surgical complications before discharge.

Follow up will be conducted at each follow-up node after surgery (1 month/3 months/6 months/12 months).

This study aims to measure the weight of patients before and after surgery, analyze the degree of weight loss based on the percentage of excess weight loss (% EWL) one year after surgery, and compare the weight loss effects of two surgical procedures.At the same time,based on relevant laboratory results,the effectiveness of two surgical procedures for treating metabolic syndrome,the incidence of postoperative nutritional complications,the incidence of surgical related complications,the quality of life one year after surgery,and weight loss were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing weight loss surgery,aged 18-65 years old
* Simple obesity with a BMI exceeding 35 or a BMI exceeding 32 combined with at least 2 metabolic syndromes
* Preoperative gastroscopy examination showed no high-risk factors for gastric cancer
* Preoperative multidisciplinary evaluation is suitable for gastric bypass or dual channel surgery
* Patients understand and accept long-term follow-up
* The patient agrees to participate in the clinical study and signs an informed consent form

Exclusion Criteria:

* The patient has type 1 diabetes
* Gastroscopy indicates active gastroduodenal ulcers within the past 2 months without treatment
* The patient has a history of chronic inflammatory bowel disease
* The patient is pregnant or has a recent pregnancy plan
* Having psychological disorders that require monitoring
* The patient has undergone weight loss surgery in the past to undergo corrective surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of excess weight loss one year after surgery (% EWL) | one year after surgery
  Percentage of excess weight loss one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xuehui Chu, Doctorate, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China